CLINICAL TRIAL: NCT01410864
Title: DuraSeal Exact Spine Sealant System Post-Approval Study
Acronym: DuraSeal PAS
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: COVDRSS0002
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Dural Sealing
Keywords: cerebrospinal fluid leaks; dural opening; dural sealing
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DuraSeal Arm: Prospective enrollment of subjects who have received DuraSeal Exact Spinal Sealant System for treatment of an intentional or incidental dural tear during spine surgery.
  Interventions: Device: DuraSeal Exact Spine Sealant System
- Control Arm: Subjects who have undergone a spinal procedure where techniques other than DuraSeal were administered for the treatment of either an intentional or incidental opening of the dura may be enrolled either prospectively or retrospectively (via medical record screening)
  Interventions: Other: Control

INTERVENTIONS:
Device: DuraSeal Exact Spine Sealant System — DuraSeal Exact Spine Sealant System will be administered to those eligible patients, to treat a dural opening.
  Groups: DuraSeal Arm
Other: Control — Devices or drugs used to seal the dura (other than DuraSeal)
  Groups: Control Arm

SUMMARY:
This is a non-randomized, post-approval study to further evaluate the rate of post-operative Cerebral Spinal Fluid (CSF) leaks in subjects who undergo a spinal procedure and receive DuraSeal Exact Spine Sealant System.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject had a spinal procedure where a dural opening (either intentional or incidental) occurred and was treated with either:

  * DuraSeal™ Exact Spine Sealant (DuraSeal™ Sealant group ONLY) OR
  * Any other method of sealing the dura with the exception of DuraSeal™ Sealant -either spinal or cranial. (Control group ONLY)
* Subject, or authorized representative, has been informed of the nature of the study and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) of the respective clinical site prior to the collection of study data.

  * Prospective subjects: Consent must be obtained within 24 hours of surgery stop time.
  * Retrospective subjects (Control group specific): IRB approval may be granted to individual sites to waive requirement for informed consent.

Exclusion Criteria:

* The investigator determines that the subject will not be able to comply with the required follow-up visits (not required if subject is being enrolled retrospectively- control group ONLY)
* Pregnant or breastfeeding females (as documented in the medical records; no testing beyond the site's standard of care is required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DuraSeal group will be patients that undergo a spinal procedure where a dural opening occurrs and is treated with DuraSeal Exact Spine Sealant System. Control group will be patients that have undergone a spinal procedure where a dural opening occurred and was treated with anything other than DuraSeal Sealant (Spine or Dural). These subjects may be enrolled retrospectively (through a chart review of past cases) or prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 924 (Actual)
Dates: Start 2011-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-operative CSF leaks | 90 days post-operative

SECONDARY OUTCOMES:
Post-operative surgical site infections | 90 days post-operative
  Deep surgical site infections as defined by the Center for Disease Control criteria.
Post-operative neurological serious adverse events | 90 days post-operative

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Phoenix, Arizona
  - Los Angeles, California
  - Sacramento, California
  - San Francisco, California
  - San Jose, California
  - Stanford, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Royal Oak, Michigan
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - East Syracuse, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Bend, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Plano, Texas
  - Charlottesville, Virginia
  - Seattle, Washington